CLINICAL TRIAL: NCT06901895
Title: Comparing Effect of Hyaluronic Acid and Lipid Coated Carbomer Gel on Dry Eyes After Phacoemulsification in Diabetic Patients
Brief Title: Comparing Effect of Hyaluronic Acid and Lipid Coated Carbomer Gel on Dry Eyes After Phacoemulsification in DP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/779
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hylorunic acid (Experimental)
  Interventions: Combination Product: Hylorunic acid
- Lipid coated carbomer gel (Active Comparator)
  Interventions: Diagnostic Test: Lipid coated carbomer gel

INTERVENTIONS:
Combination Product: Hylorunic acid — Hylorunic acid (hylo) eye drop is prescribed and check the curative effect after phacoemulsification after 2nd and 4th week.
  Arms: Hylorunic acid
Diagnostic Test: Lipid coated carbomer gel — Lipid coated carbomer gel (visole)is prescribed and check yhe curative effect after phacoemulsification in diabetic patients post operatively in 2nd and 4th week.
  Arms: Lipid coated carbomer gel

SUMMARY:
In this study we compare the curative effect of two lubricants Hylorunic acid and visol gel on dry eyes after phacoemulsification in diabetic patients. We check the tear film before operation and check post operate after 2nd week and 4th week of surgery. Its a hospital based study .

ELIGIBILITY:
Inclusion Criteria:

* Patients who have acute dry eye condition before phacoemulsification cataract surgery.

Exclusion Criteria:

* Patients who have chronic dry eye condition before phacoemulsification cataract surgery.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Schirmer test | 12 Months
  The Schirmer's test, also known as the Schirmer tear test, is a medical test used to assess tear production, particularly when a person experiences dry eyes or excessive tearing, by measuring how much a filter paper strip gets wet by tears in the lower eyelid
Tear Break up Test | 12 months
  The Tear Breakup Time (TBUT) test, also known as the Tear Film Breakup Time (TFBUT) test, assesses tear film stability by measuring the time it takes for dry spots to appear on the cornea after a blink, indicating potential dry eye

CONTACTS AND LOCATIONS:
Locations (1):
- Shaheen welfare hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No